CLINICAL TRIAL: NCT03874325
Title: A Phase II Trial With Safety Run-in of Neoadjuvant Therapy With an Aromatase Inhibitor in Combination With Durvalumab (MEDI4736) in Postmenopausal Patients With Hormone-Receptor-Positive Breast Cancer
Brief Title: Aromatase Inhibitor and Durvalumab in Postmenopausal Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lost funding
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19803; ESR-17-13182 (Other: AstraZeneca)
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Results first posted 2022-01-11 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer; Hormone Receptor Positive Tumor
Keywords: HR+
MeSH Terms: conditions — Breast Neoplasms | interventions — durvalumab; Anastrozole; Letrozole; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Safety Run In: Durvalumab + Aromatase Inhibitor (Experimental): Participants will be administered 1500 mg Durvalumab intravenously every 4 weeks for 6 cycles. Participants will also take standard of care 1 mg anastrozole daily by mouth for 6 months. Letrozole 2.5 mg or exemastane 25 mg may be substituted for anastrozole if an intolerance to anastrozole is exhibited. Six participants will be enrolled in the safety run in stage. If 1 or fewer of six participants have a DLT, expansion stage will open to enrollment.
  Interventions: Drug: Durvalumab; Drug: Anastrozole 1mg; Drug: Letrozole 2.5mg; Drug: Exemestane 25 MG
- Expansion: Durvalumab + Aromatase Inhibitor (Experimental): Participants will be administered 1500 mg Durvalumab intravenously every 4 weeks for 6 cycles. Participants will also take standard of care 1 mg anastrozole daily by mouth for 6 months. Letrozole 2.5 mg or exemastane 25 mg may be substituted for anastrozole if an intolerance to anastrozole is exhibited.
  Interventions: Drug: Durvalumab; Drug: Anastrozole 1mg; Drug: Letrozole 2.5mg; Drug: Exemestane 25 MG

INTERVENTIONS:
Drug: Durvalumab — 1500 mg Durvalumab will be administered intravenously every 4 weeks for 6 months.
  Other Names: MEDI4736
Drug: Anastrozole 1mg — Participants will self administer 1 mg anastrozole by mouth daily for 6 months.
  Other Names: Arimidex
Drug: Letrozole 2.5mg — Participants intolerant to anastrozole will self administer 2.5 mg letrozole by mouth daily for 6 months. Exemestane may be substituted.
  Other Names: Femara
Drug: Exemestane 25 MG — Participants intolerant to anastrozole will self administer 25 mg exemestane by mouth daily for 6 months. Letrozole may be substituted.
  Other Names: Aromasin

SUMMARY:
This study is to find out if an investigational drug called Durvalumab (MEDI4736) given together with a standard of care aromatase inhibitor drug can help people with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Postmenopausal, defined as meeting criteria per protocol.
* Clinical T2-T4c, any N, MO by American Joint Committee on Cancer staging, 8th edition, with the goal being definitive surgery after completion of neoadjuvant therapy. Tumor is palpable and its size can be measured bidimensionally by tape, ruler or caliper technique. Largest tumor diameter over 2.0 cm.
* Pathologic confirmation of invasive breast cancer that is estrogen receptor (ER) positive as defined in the protocol.
* Invasive breast cancer is Human Epidermal Growth Factor Receptor 2 (HER2) negative as defined in the protocol protocol.
* Documentation of mammogram and ultrasound [including ductal carcinoma in situ (DCIS) and invasive cancer] of the diseased breast performed within 60 days prior to enrollment. Mammograms for the unaffected contralateral breast is required within 12 months prior to enrollment.
* Adequate organ and marrow function, as defined in the protocol.
* Participants must be willing to undergo a research biopsy at baseline and after one cycle of treatment and to provide tissue obtained at surgery for biomarker and correlative studies.
* Participants must be willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* If taking herbal or natural remedies that may have immune modulatory effects, participants must be willing to discontinue use prior to first dose of durvalumab.
* Body weight over 30 kg.

Exclusion Criteria:

* Participation in another clinical study with an investigational product during the last 4 weeks.
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow up period of an interventional study.
* Inflammatory breast cancer defined as clinically significant erythema of the breast and/or documented dermal lymphatic invasion (not direct skin invasion by tumor or peau d'orange without erythema).
* An excisional biopsy of this breast cancer. Hormone replacement therapy of any type, megestrol acetate, or raloxifene within one week prior to registration.
* Surgical axillary staging procedure prior to study entry. Note: Fine needle aspiration (FNA) or core needle biopsy of axillary node is permitted.
* Treatment for this cancer including surgery, radiation therapy, chemotherapy, biotherapy, hormonal therapy or investigational agent prior to study entry.
* Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab
* History of another primary malignancy except for malignancy treated with curative intent and with no known active disease ≥ 5 years or adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease or adequately treated carcinoma in situ without evidence of disease e.g., cervical cancer in situ.
* History of ipsilateral invasive breast cancer regardless of treatment or ipsilateral ductal carcinoma in situ (DCIS) treated with radiotherapy or endocrine therapy or contralateral invasive breast cancer at any time.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab, with the exceptions of intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra-articular injection); systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid; or steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). Some exceptions apply.
* History of primary immunodeficiency.
* History of allogeneic organ transplant.
* Known allergy or history of hypersensitivity to durvalumab, or any excipient.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses, , or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.
* Known active infection including tuberculosis, hepatitis B, hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved hepatitis B infection are eligible. Patients positive for hepatitis C antibody are eligible only if polymerase chain reaction is negative for hepatitis C RNA. Note: This is applied only to patients with known infection. Screening tests for TB, hepatitis B and C, or HIV are not required.
* Receipt of live attenuated vaccination within 30 days prior to receiving durvalumab. Note: Patients, if enrolled, should not receive live vaccine while receiving durvalumab and up to 30 days after the last dose of durvalumab.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.
* Participants with uncontrolled seizures.
* Participants with multi-centric breast cancer (defined as more than one lesion is invasive breast cancer in the same breast separated by ≥ 2 cm of normal breast tissue).
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of investigational product.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 17 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2021-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hung Khong, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Safety Run In: Durvalumab + Aromatase Inhibitor | Expansion: Durvalumab + Aromatase Inhibitor
Started | 17 | 0
Completed | 17 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study terminated early and did not go beyond Safety run in
Groups:
- Safety Run In: Durvalumab + Aromatase Inhibitor: Study terminated early and did not move beyond safety run in.
  Participants administered 1500 mg Durvalumab intravenously every 4 weeks for 6 cycles. Participants took standard of care 1 mg anastrozole daily by mouth for 6 months. Letrozole 2.5 mg or exemastane 25 mg may be substituted for anastrozole if an intolerance to anastrozole is exhibited. Six participants will be enrolled in the safety run in stage. If 1 or fewer of six participants have a DLT, expansion stage will open to enrollment.
  Durvalumab: 1500 mg Durvalumab will be administered intravenously every 4 weeks for 6 months.
  Anastrozole 1mg: Participants will self administer 1 mg anastrozole by mouth daily for 6 months.
  Letrozole 2.5mg: Participants intolerant to anastrozole will self administer 2.5 mg letrozole by mouth daily for 6 months. Exemestane may be substituted.
  Exemestane 25 MG: Participants intolerant to anastrozole will self administer 25 mg exemestane by mouth daily for 6 months. Letrozole may be substituted.
Arm/Group | Safety Run In: Durvalumab + Aromatase Inhibitor
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Rate of Modified Preoperative Endocrine Prognostic Index (mPEPI) Score of 0
Description: Modified preoperative endocrine prognostic index (mPEPI) of 0. Total PEPI score assigned to each patient is the sum of the risk points derived from the pathological (pT) stage, lymph node (pN) stage, Ki67 level, and estrogen receptor (ER) status of the surgical specimen. A hazard ratio (HR) in the range of 1-2 receives one risk point; a HR in the 2-2.5 range, two risk points; a HR greater than 2.5, three risk points.
  mPEPI score of 0 indicates a tumor size of 5 cm or less, negative lymph nodes, and Ki67 (proliferation index) of less than or equal to 2.7%. Drug combination will be determined to be efficacious if 7 or more participants achieve an mPEPI of 0.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Safety Run In: Durvalumab + Aromatase Inhibitor
Number analyzed (Participants) | 17
percentage of participants | 17.65 [3.8 to 43.43]

2. Secondary Outcome: Clinical Complete Response (CR)
Description: Clinical Complete response: Palpable lesion(s) identified at baseline are no longer palpable and there are no new lesion(s) or other signs of disease progression.
Time Frame: 6 months
Measure: Number; unit: percentage of patients
Arm/Group | Safety Run In: Durvalumab + Aromatase Inhibitor
Number analyzed (Participants) | 17
percentage of patients | 58.8

3. Secondary Outcome: Clinical Partial Response (PR)
Description: Clinical Partial response: A reduction in the product of the two largest perpendicular diameters of the primary tumor by 50% or more.
Time Frame: 6 months
Measure: Number; unit: percentage of patients
Arm/Group | Safety Run In: Durvalumab + Aromatase Inhibitor
Number analyzed (Participants) | 17
percentage of patients | 41.2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first study drug administration to 90 days post last dose of study treatment. Study terminated prematurely, adverse events were collected for 20 months
Arm/Group | Safety Run In: Durvalumab + Aromatase Inhibitor
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 2/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Run In: Durvalumab + Aromatase Inhibitor (N=17)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Vomitting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Run In: Durvalumab + Aromatase Inhibitor (N=17)
Fatigue (General disorders) | 12 (17)
Pain (General disorders) | 4 (7)
Edema limbs (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (3)
Chills (General disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Neck edema (General disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (13)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Intraoperative breast injury (Injury, poisoning and procedural complications) | 2 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Headache (Nervous system disorders) | 8 (9)
Dizziness (Nervous system disorders) | 4 (5)
Dysgeusia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (9)
Diarrhea (Gastrointestinal disorders) | 5 (7)
Constipation (Gastrointestinal disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Dental caries (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 (3)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (2)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flashes (Vascular disorders) | 8 (9)
Hypotension (Vascular disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 5 (5)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 4 (5)
Hyperthyroidism (Endocrine disorders) | 2 (2)
Endocrine disorders - Other (Endocrine disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin infection (Infections and infestations) | 2 (2)
Herpes simplex reactivation (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Allergic reaction (Immune system disorders) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1)
Gallbladder pain (Hepatobiliary disorders) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/25/NCT03874325/Prot_SAP_000.pdf